CLINICAL TRIAL: NCT02009917
Title: Application of Indicator Amino Acid Oxidation Technique to Determine Non-essential Amino Acids/Nitrogen Requirements in Adult Humans
Brief Title: Non- Essential Amino Acid Requirements and Metabolism in Humans
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: Ajinomoto Co., Inc. (Industry)
Responsible Party: Principal Investigator, Rajavel Elango, PhD, Principle Investigator, University of British Columbia
Other Study IDs: H12-01683
Record Dates: First submitted 2013-12-09; First posted 2013-12-12 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Healthy Adult Males
Keywords: Indicator Amino Acid Oxidation; Non essential Amino acids; Protein; Amino acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Breath and urine samples
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Protein is a major structural component of all cells in the body. The nutritional importance of protein is because of their amino acids. 9 are called essential and 11 are called non-essential, based on whether we need to get them from diet. This classification is based on studies done using older techniques. Recent studies suggest that these so called non-essential amino acids play important roles in our body's health. For the first time, this proposal defines an experimental design to examine non- essential amino acid/nitrogen requirements and metabolism in humans using the Indicator Amino Acid Oxidation (IAAO) technique.

The objective of the current study is to examine the application of IAAO technique to determine the non-essential amino acid/nitrogen requirement in adult humans.

ELIGIBILITY:
Inclusion Criteria:

* 20-40 years of age
* Male
* Classified as normal body weight based on body mass index (BMI) 18.5-25kg/m2
* Free of any concurrent illness

Exclusion Criteria:

* Men not in good health or have a metabolic, neurological, genetic or immune disorder including diabetes and hypertension
* Men who are classified as underweight(<18.5kg/m2), overweight(25-30kg/m2) or obese (>30kg/m2) using the BMI classification)
* Men who are allergic to milk, eggs and egg protein

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Physiologically Healthy Adult males, 20-40 years of age
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2013-10; Primary Completion 2015-01 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
13 Carbon dioxide production | 8 hours (1study day)
  Urine and breath samples will be collected to measure the rate of oxidation of expired breath and flux by enrichment of urine.

CONTACTS AND LOCATIONS:
Overall Officials: Rajavel Elango, Ph.D, Principal Investigator — University of British Columbia
Locations (1):
- Child and Family Research Institute, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Cooper L, Ball RO, Pencharz PB, Sakai R, Elango R. Dispensable Amino Acids, except Glutamine and Proline, Are Ideal Nitrogen Sources for Protein Synthesis in the Presence of Adequate Indispensable Amino Acids in Adult Men. J Nutr. 2020 Sep 1;150(9):2398-2404. doi: 10.1093/jn/nxaa180. PMID 32879983